CLINICAL TRIAL: NCT00912236
Title: Evaluation of High-Density Lipoprotein in Obesity Study
Status: Terminated | Type: Observational
Why Stopped: Investigator left institution
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 09-302
Record Dates: First submitted 2009-05-20; First posted 2009-06-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Obesity; HDL; HDL functionality
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: BMI 20-25 kg/m2
- 2: BMI > 30 kg/m2 with low TG (<150) and normal HDL (>50 for females, >40 for males)
- 3: BMI > 30 kg/m2 with high TG (>150) and low HDL (<50 for females, <40 for males)

SUMMARY:
Obesity is associated with an impaired functioning HDL (good cholesterol) resulting in an acceleration in the development of atherosclerosis. This study will evaluate HDL functionality in patients with BMI (Body Mass Index) 20 - 25 and BMI >30

DETAILED DESCRIPTION:
This study will determine if the protective function of high-density lipoprotein (HDL) is impaired in obese patients and will help to enhance cardiovascular risk prediction. Carotid intima-media thickness (cIMT) will be captured as a means of assessing early vascular changes associated with low HDL levels in obesity. A novel measurement for clinical correlation has also been introduced called carotid extra-medial thickness (cEMT) which will be compared to cIMT in this obese population.

ELIGIBILITY:
Inclusion Criteria:

* Group 1:

  * Age 20-80
  * English speaking
  * BMI 20-25 kg/m2
* Group 2:

  * Age 20-80
  * English speaking
  * BMI > 30 kg/m2
  * TG > 150 and
  * HDL > 50 (females) >40 (Males)
* Group 3:

  * Age 20-80
  * English speaking
  * BMI > 30 kg/m2
  * TG > 150 and
  * HDL < 50 (females) < 40 (males)

Exclusion Criteria:

* Self-reported history of:

  * Diabetes mellitus
  * Any previous lipid therapy within the last three months
  * Macrovascular events including TIA, stroke, myocardial infarction, heart failure, claudication, or known peripheral vascular disease
  * Current pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from Cleveland Clinic outpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine whether the functional activity of HDL is impaired in the setting of obesity | Within 2 weeks of enrollment

SECONDARY OUTCOMES:
To determine whether HDL is more susceptible to oxidative modification ex-vivo in obese patients by mass spectrometry | Within 2 weeks of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, MBBS, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No